CLINICAL TRIAL: NCT02095730
Title: Study of Safety and Efficacy of Photochemically Induced Collagen Cross-Linking at an Irradiance of 18 mW/cm2 as Constant or Pulsed Treatment in Eyes With Unstable Corneas Due to Keratoconus, Ectasia, or Post-Incisional Refractive Surgery
Brief Title: Corneal Cross-Linking Comparing Variables
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Crowd Health Research, LTD (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CXL-CHR 1
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Unstable Corneas
Keywords: crosslinking; cornea; keratoconus; ectasia; irradiance; riboflavin
MeSH Terms: conditions — Corneal Diseases; Keratoconus; Dilatation, Pathologic | interventions — Riboflavin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Epi-On Continuous (Active Comparator): Continuous beam of UV light treating cornea with surface epithelium present
  Interventions: Drug: Epithelium-On Riboflavin; Device: UV Light - Continuous Beam
- Epi-Off Continuous (Active Comparator): Continuous beam of UV light treating cornea without surface epithelium present
  Interventions: Drug: Epithelium-Off Riboflavin; Device: UV Light - Continuous Beam
- Epi-On Pulsed (Active Comparator): Pulsed beam of UV light treating cornea with surface epithelium present
  Interventions: Drug: Epithelium-On Riboflavin; Device: UV Pulsed Beam
- Epi-Off Pulsed (Active Comparator): Pulsed beam of UV light treating cornea without surface epithelium present
  Interventions: Drug: Epithelium-Off Riboflavin; Device: UV Pulsed Beam

INTERVENTIONS:
Drug: Epithelium-On Riboflavin — Riboflavin 0.1% Phosphate Sodium solution with Benzalkonium Chloride Preservative
  Other Names: Vitamin B2
  Arms: Epi-On Continuous; Epi-On Pulsed
Drug: Epithelium-Off Riboflavin — Riboflavin 0.1% Phosphate Sodium solution
  Other Names: Vitamin B2
  Arms: Epi-Off Continuous; Epi-Off Pulsed
Device: UV Light - Continuous Beam — 5 minutes of constant UV exposure to saturated cornea
  Other Names: Peschke Vario CCL-365 UV system
  Arms: Epi-Off Continuous; Epi-On Continuous
Device: UV Pulsed Beam — 5 minutes of UV exposure to saturated cornea, alternating 1 minute of treatment with 1 minute rest for a total time of 10 minutes
  Other Names: Peschke Vario CCL-365 UV system
  Arms: Epi-Off Pulsed; Epi-On Pulsed

SUMMARY:
The purpose of this study is to evaluate the Safety and Efficacy of Corneal Cross Linking in a Continuous Beam versus Pulsed Treatments across epithelium on and epithelium off surfaces.

ELIGIBILITY:
Inclusion Criteria Keratoconus:

* 12 years of age or older
* Having a clinical diagnosis of progressive keratoconus consistent with:

  1. An increase of ≥ 1.00 D in the steepest keratometry value
  2. An increase of ≥ 1.00 D in astigmatism manifest refraction
  3. A myopic shift (decrease in the spherical equivalent) of ≥ 0.50 D on subjective manifest refraction
* Presence of central or inferior steepening on the topography map.
* Axial topography consistent with keratoconus
* Steepest keratometry (Kmax) value ≥ 47.00 D
* Signed written informed consent
* Willingness and ability to comply with schedule for follow-up visits
* Contact lens removal prior to evaluation and treatment

Inclusion Criteria Post-Surgical Ectasia:

* History of having undergone a keratorefractive procedure and:

  1. Steepening by topography
  2. Thinning of cornea
  3. Shift in the position of thinnest portion of cornea
  4. Change in refraction with increasing myopia
  5. Development of myopic astigmatism
  6. Development of irregular astigmatism
  7. Loss of Best Spectacle Corrected Visual Acuity
* At least two of the above criteria must be present.

Inclusion Criteria Intacts:

* Should the patient have undergone prior Intacs or other intra-corneal ring segment surgery for keratoconus or post-surgical ectasia at least 6 months prior, and is also experiencing at least two of the above ectasia symptoms, they can be included in the study.

  1. These patients would have the choice of ring explant before Cross-Linking.
  2. Cross-Linking may still be performed if the patient wishes to retain the rings.
* Should a patient's situation due to factors such as significantly high myopia or astigmatism should warrant simultaneous placement of Intacs and cross-linking in the investigators opinion, then this option can be offered to the patient. Such interventions would be tracked as a different arm of the study.

Inclusion Criteria RK/AK Fluctuation:

* History of having undergone radial keratotomy (RK) and or astigmatic keratotomy (AK) surgery.
* Expressing complaints about difficulties due to vision changing during the same day.
* A difference in their Manifest Refraction (MRx) of greater than 0.75 D measured on the same day, at least 6 hours apart.
* Intacs surgery will not be considered in patients with RK/AK.

Exclusion Criteria:

* Eyes classified as either normal, atypical normal,
* Corneal pachymetry ≤ 350 microns at the thinnest point measured by Orbscan, Pentacam, or ultrasound in the eye to be treated
* A history of chemical injury or delayed epithelial healing in the eye to be treated.
* A known sensitivity to study medications
* Patients with significant nystagmus or any other condition that would prevent a steady gaze during the treatment
* Inability to cooperate with diagnostic tests.
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.
* Taking Vitamin C (ascorbic acid) supplements within 1 week of the cross-linking treatment.
* Patients who are unable to remain comfortable and stable, and tolerate a lid speculum for the appointed period of time for the procedure.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 2 years
  Uncorrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Tanchel, MD, Principal Investigator — Liberty Laser Eye Center
Locations (16):
- United States (16):
  - LaserVue Eye, Santa Rosa, California
  - Icon Lasik, Denver, Colorado
  - Gulani Vision Institute, Jacksonville, Florida
  - Eye Consultants of Atlanta, Atlanta, Georgia
  - Midwest Center for Sight, Des Plaines, Illinois
  - Bond Eye Associates, Pekin, Illinois
  - Discover Vision Center, Leawood, Kansas
  - Southern Eye Center, Hattiesburg, Mississippi
  - Mercy Clinic Eye Specialists, Springfield, Missouri
  - LASIK of Nevada, Las Vegas, Nevada
  - James Lewis MD PC, Elkins Park, Pennsylvania
  - Memorial Eye Institute, Harrisburg, Pennsylvania
  - Carolina Eye Care, Mt. Pleasant, South Carolina
  - Loden Vision Centers, Goodlettsville, Tennessee
  - Parkhurst NuVision, San Antonio, Texas
  - Liberty Laser Eye Center, Vienna, Virginia